CLINICAL TRIAL: NCT00365443
Title: Proprietary Information - Exploratory (Non-Confirmatory) Trial
Brief Title: Broad Spectrum HPV Vaccine Tolerability, Immunogenicity, and Efficacy Study (V502-003)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V502-003; 2006_503
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Cervical Cancer; Condylomata Acuminata
Keywords: anogenital warts; premalignancy; HPV; Human papillomavirus
MeSH Terms: conditions — Uterine Cervical Neoplasms; Condylomata Acuminata

INTERVENTIONS:
Biological: V502

SUMMARY:
This study is to evaluate an investigational vaccine with the following objectives: (1) To demonstrate prevention of cervical, vulvar, and vaginal cancers and related precancers, external genital lesions, and persistent infection caused by the HPV types in the study vaccine, (2) To demonstrate that the vaccine is well-tolerated in women, (3) To evaluate vaccine immune responses in women.

This is an early phase trial and some specific protocol information is proprietary and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* Female, between the ages of 16 and 26

Exclusion Criteria:

* History of an abnormal PAP test or abnormal cervical biopsy result
* History of external genital/vaginal warts
* History of positive HPV test
* Currently a user of any illegal drugs or an alcohol abuser
* Are pregnant
* Currently enrolled in another clinical trial
* Currently has or has a history of certain medical conditions or is currently taking or has taken certain medications (details will be discussed at the time of consent).

Ages: 16 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10

PRIMARY OUTCOMES:
Proprietary Information - Exploratory (Non-Confirmatory) Trial

SECONDARY OUTCOMES:
Proprietary Information - Exploratory (Non-Confirmatory) Trial

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC